CLINICAL TRIAL: NCT00183131
Title: Internet Screening and Brief Intervention for Hazardous Drinking in College Students: A Pilot Study
Brief Title: The iHealth Study in College Students
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Boston University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIAAASAI013759; P60AA013759 (NIH); NIH P60 AA013759
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2007-12

CONDITIONS: Alcohol Abuse; Alcohol Dependence; Unhealthy Alcohol Use; Risky Alcohol Consumption Amounts; Hazardous Alcohol Use
Keywords: Alcohol; Alcohol abuse; Alcohol dependence; Alcohol consumption; Unhealthy alcohol use; Screening; Brief Intervention; Effectiveness; Electronic intervention; Web-based intervention; College students
MeSH Terms: conditions — Alcoholism; Alcohol Drinking

INTERVENTIONS:
Behavioral: Brief Personalized Feedback

SUMMARY:
The objective of this project was to test the feasibility of electronic mail recruitment and web screening for hazardous drinking, to compare different approaches to encouraging screening, and to estimate the effects of minimal and more extensive feedback in preparation for a future alcohol web-based brief intervention study

DETAILED DESCRIPTION:
This pilot study aims to test the feasibility of electronic mail recruitment and web screening for alcohol problems, to compare different approaches to encouraging screening, and to estimate the effects of minimal and more extensive feedback in preparation for a future alcohol web-based brief intervention study. To do so, 4300 freshman adult college students will be randomized to receive an electronic mail request to complete a web alcohol screening test using an alcohol-specific or a general wellness approach. The primary outcome is the proportion of respondents who complete alcohol screening. Additional outcomes include readiness to change drinking, help-seeking, alcohol consumption and consequences. The results of this pilot study will provide information useful to 1) colleges deciding how best to implement universal screening for hazardous alcohol use, and 2) in the preparation of a larger study of web-based screening and brief intervention for hazardous drinking in college students.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Full time student
* College freshman

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4300
Dates: Start 2004-10; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Change in the number of times a subject exceeded per occasion limits
Drinking risky amounts
Heavy episodic drinking
Drinks per day
Hazardous drinking

SECONDARY OUTCOMES:
Abstinence
Readiness to change alcohol use
Help-seeking
Alcohol consequences

CONTACTS AND LOCATIONS:
Overall Officials: Richard Saitz, M.D., M.P.H., Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Saitz R, Helmuth ED, Aromaa SE, Guard A, Belanger M, Rosenbloom DL. Web-based screening and brief intervention for the spectrum of alcohol problems. Prev Med. 2004 Nov;39(5):969-75. doi: 10.1016/j.ypmed.2004.04.011. PMID 15475031
- See also: AlcoholScreening.org is an anonymous, free online self-screening service to assess an individual's alcohol consumption and its consequences. — http://www.alcoholscreening.org